CLINICAL TRIAL: NCT06442423
Title: Safety, Feasibility, and Tolerability of Psilocybin Treatment for Individuals With Functional Impairment Related to Mood, Anxiety, Trauma and/or Addiction Symptoms: An Open-label Proof-of-concept Study
Brief Title: Open-Label Psilocybin Study in Transdiagnostic Population
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Principal Investigator, Benjamin Kelmendi, MD, Assistant Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000037785
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Transdiagnostic; Depression - Major Depressive Disorder; Anxiety; PTSD Symptoms; PTSD; Substance Use; Substance Use Disorder (SUD); OCD
Keywords: depression; anxiety; substance use; addiction; PTSD; OCD; psilocybin; psychedelic
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Depression; Behavior, Addictive | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: We will employ an unblinded, open-label study where all participants will be given one dose of oral psilocybin 25mg. We will also have follow-up visits at 1, 4, and 6 weeks and an optional long-term follow-up at 3, 6, and 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Other): Psilocybin will be administered in an opaque, size 2 gelatin capsule with approximately 180 ml of water to be orally ingested at Visit 5. The dose of psilocybin will be 25 mg.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin will be administered in an opaque, size 2 gelatin capsule with approximately 180 ml of water to be orally ingested at Visit 5. The dose of psilocybin will be 25 mg.This is an open-label clinical trial with a single treatment arm. This is an open-label clinical trial with no blinding.

SUMMARY:
The primary objective of this study is to investigate the safety, feasibility, and tolerability of psilocybin treatment in individuals with functional impairment due to psychiatric symptoms. The secondary objective of this study is to determine whether individuals with functional impairments due to psychiatric symptoms will experience statistically significant symptom reduction and functional improvement from baseline symptom measurements (Visit 3) to 1-week (Visit 7), 4-weeks (Visit 8), and 6-weeks (Visit 9) post dosing. The investigators will recruit individuals with mood, anxiety, trauma, addictive, or related symptomatology, and who have functional impairment associated with these symptoms. A DSM-5 diagnosis is not required (nor is it an exclusion). The investigators will allow for comorbidity and only exclude based on psychological and physiological safety considerations. Critically, this approach will allow us to assess the tolerability of our interventions in individuals who would typically be excluded from efficacy studies due to various comorbid DSM-5 conditions.

The investigators will employ an open-label study where participants will be given one dose of oral psilocybin 25mg. The investigators will also have follow-up visits at 1, 4, and 6 weeks and an optional long-term follow-up at 3, 6, and 12 months.

DETAILED DESCRIPTION:
In this Phase 1b proof-of-concept clinical trial, the investigators aim to investigate the safety, feasibility, and tolerability of treatment of oral psilocybin in participants with functional impairment due to depressive, anxiety, trauma addictive, or other psychiatric symptomatology, allowing for comorbidity and diagnostic complexity to mirror potential real-world clinical scenarios. Secondarily, The investigators will assess improvement in functional status and symptomatology.

The investigators will employ an open-label study design, with participants receiving one dose of oral psilocybin. This is an open-label clinical trial with a single treatment arm and no blinding. All participants will receive 25 mg of oral psilocybin. All dosing will be accompanied by non-directive support before, during, and after treatment sessions.The rationale for conducting this study lies in recognizing that the narrow inclusion and exclusion criteria commonly employed in clinical trials may raise issues of external validity. While previous research has predominantly focused on specific diagnostic categories, our study aims to address these limitations by exploring the safety, feasibility, and tolerability of psilocybin in a heterogeneous population.

This study also recognizes the importance of symptom-related functional impairment as a cross-cutting construct relevant to all diagnostic categories.This is a Phase 1b open-label clinical trial to determine the feasibility, tolerability and safety of psilocybin to reduce psychiatric symptoms in participants experiencing functional impairment. Participants will receive one dose of oral psilocybin (25mg). Follow-up visits for assessments and measures at 1-week, 4-week, and 6-week post psilocybin dosing. Long-term follow-up visits assessments and measures for participants who consent to long-term follow-up (reassessments of study measures) for 3-month, 6-month, and 12-month post dosing.

Psilocybin (4-hydroxy-N,N-dimethyltryptamine) occurs in nature in many species of mushrooms, including the genera Psilocybe, Conocybe, Gymnopilus, Panaeolus, and Strophparia. Its chemical formula is C12H17N2O4P. Psilocybin is a potent agonist at 5-HT2A/C receptors; potency of binding by related compounds to these receptors correlates with human potency as hallucinogens. Psilocybin is currently a Schedule I substance. Psilocybin will be orally administered in this study. Psilocybin will be administered in an opaque, size 2 gelatin capsule with approximately 180 ml of water to be orally ingested at Visit 5. The dose of psilocybin will be 25 mg.

Descriptives for all safety measures (e.g., C-SSRS total and subscale scores, vitals, documented adverse events) will be compiled at all assessment intervals. Classification of adverse events will follow institute and regulatory body guidelines. Subsequent summary descriptives may focus on safety indices surrounding the dosing session and 1-week, 4 weeks, and 6-weeks after dosing. In addition, The investigators will perform descriptives and non-parametric analysis screen failure rates (including analysis of ineligibility), drop out rates pre and post dosing to determine feasibility and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. At least one psychiatric symptom causing functional impairment over the past 30 days as established by a trained rater on the DIAMOND (at least "mild" impairment) and/or the WHODAS-2.0 12-item (a raw score of >16) - assessment instruments indexing health and disability.
2. English fluency - able to understand the process of consent and the risk and benefits associated with the study, and able to provide written (signed and dated) informed consent form.
3. Agree to set up safe transportation after leaving the site following the dosing session. Acceptable arrangements include: arranging for a friend/family member to drive them home, pick them up and escort them home; if the participant is unable to arrange for a friend/family member to escort them home, the study staff will arrange private transportation and follow up with the participant to ensure that they arrived at their destination.
4. Must be able to identify a physician/treater that can be contacted to further assure that it is safe for the subject to participate and agree to sign a medical release for the investigators to communicate directly with this outside provider to confirm treatment and medical history via phone and/or email.
5. Ability to orally ingest pills for psilocybin dosing visit.
6. Must provide an adult contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the PI and/or study personnel in the event of an emergency, and who can provide transportation for study visits if necessary and independently comment on any changes in the participant's mood or behavior after the administration of psilocybin. Be medically stable (no medical issues based on physical exam, labs and medical evaluation) as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an ECG, and routine blood and urinalysis laboratory tests (see section 6.3.4 for labs). Must also demonstrate decisional capacity based on clinical assessment ensuring the participant can understand, appreciate, and reason through the study's purpose, procedures, and associated risks, as well as tolerate the potential effects of the study medication.
7. Be psychologically stable: Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least one month prior to screening and is expected to remain stable during participation in the study (up to 4-weeks post-dosing).
8. If participant is of childbearing potential, must agree to use adequate birth control and not attempt to become pregnant during study up to 4 weeks post dosing session (see Section 6.3.3).

If participant is of childbearing potential, must have a negative urine pregnancy test at study entry and prior to the dosing session. Participants who are FOCBP must not plan to become pregnant or donate eggs, starting at least 1 month before receiving the trial intervention and for at least 1 week after the final follow-up visit.

A FOCBP is defined as a female who is considered fertile following menarche and until becoming postmenopausal, unless permanently sterile (see below).

Females in the following categories are not considered FOCBP:

* Premenarchal.
* Premenopausal with 1 of the following:

  1. Documented hysterectomy or bilateral salpingectomy/tubal occlusion/oophorectomy.
  2. Postmenopausal.
* A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Females receiving hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use 1 of the nonhormonal, highly effective contraception methods if they wish to continue their HRT during the trial.

Exclusion Criteria:

Psychiatric Exclusion Criteria:

1. Personal history of a primary psychotic disorder (e.g., schizophrenia, delusional disorder, schizoaffective disorder) or Bipolar I disorder, or at least one first-degree relative with a diagnosis of primary psychotic disorder (e.g., schizophrenia, delusional disorder, schizoaffective disorder) or Bipolar I disorder.
2. Active suicidal intent or suicidal or non-suicidal self-injurious behaviors, as defined by a "yes" response to question 4 on C-SSRS within the past 6 months at screening or prior to dosing (Active Suicidal Ideation with Some Intent to Act, with or without Specific Plan).
3. Use of a classic psychedelic (i.e., LSD, psilocybin, DMT, mescaline) within the 3 months prior to enrollment (not including microdosing).
4. Use of ketamine within the past month at Screening.
5. History of regular and frequent use of a classic psychedelic (more than 10 times per year) in a structured, intentional setting over the past 10 years. Structured use refers to participation in organized retreats, ceremonies, or church services. Microdosing is not included.
6. History of Other Hallucinogen Use Disorder.
7. History of intolerance to drugs known significantly to alter perception (i.e., psilocybin, LSD, salvinorium A, mescaline).
8. Patients taking 5-hydroxytryptophan or St. John's Wort
9. A positive breathalyzer test
10. A positive urine toxicology screening, which detects the standard panel of five drugs (marijuana, cocaine, opioids/opiates, amphetamines, and phencyclidine (PCP)), as well as benzodiazepines, 3,4-methylenedioxymethamphetamine (MDMA). If a participant tests positive for any of these substances, the PI may request a retest during the screening phase. The exceptions to the exclusion are prescribed opioid pain medication and benzodiazepines, or over-the-counter non-narcotic pain medication. If a participant is prescribed benzodiazepines, the participant will be asked to refrain from taking on the day of the psilocybin dosing session. Additionally, participants will not be excluded from the study based on the use of cannabis. However, they will be instructed to refrain from use of cannabis on the day before, day of, and day following the drug administration session. Participants whose primary clinical presenting issue is substance use-related will not be excluded based on a positive test at screening but will be expected to adhere to the dosing day drug test produces (outlined in section 6.3.6).
11. Changes to psychotropic medication and/or dosages within the past 3 months.
12. Current or recent (within 2 weeks of enrollment) prescription of MAOI, Lithium, and/or methadone use.
13. Has a psychiatric condition that precludes the establishment of therapeutic rapport as evidenced by long-term patterns of unstable relationships, a history of significant stress- related paranoia, or identity disturbances.
14. Use of any other investigational drugs within 30 days prior to Screening.
15. Allergy to gelatin.

General Medical/Laboratory Exclusion Criteria:

1. Hypertension at screening is defined as: systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg, on the lowest of three measurements.
2. History of cardiovascular disease, including but not limited to clinically significant coronary artery disease, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, angina pectoris, coronary artery bypass graft or artificial heart valve, stroke, transient ischemic attack, or any clinically significant arrhythmia.
3. Any clinically significant abnormal electrocardiogram (ECG) finding, such as findings suggestive of ischemia or infarct, complete bundle branch block, atrial fibrillation or other symptomatic arrhythmias, or predominantly non-sinus rhythm, at Screening.
4. Resting QT interval with Fridericia's correction (QTcF) ≥ 450 msec (male) or ≥ 470 msec

   a. (female) at Screening, or inability to determine QTcF interval.
5. Presence of risk factors for torsades de pointes, including: long QT syndrome, uncontrolled hypokalemia or hypomagnesemia, history of cardiac failure, history of clinically significant/symptomatic bradycardia, family history of idiopathic sudden death or congenital long QT syndrome, or concomitant use of a torsadogenic medication.
6. Moderate-to-severe hepatic impairment, defined as a Child-Pugh score ≥ 5, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x the upper limit of normal (ULN), or bilirubin > 1.5 x ULN, unless this is attributable to Gilbert's syndrome
7. Use of vasoconstrictive medications (i.e. sumatriptan, pseudoephedrine, midodrine) within 5 half-lives of test days and use of steroids or certain other immunomodulatory agents (i.e. azathioprine) in the past 2 weeks.
8. Moderate-to-severe renal impairment, defined as an estimated glomerular filtration rate of < 50 mL/min/1.73 m2 at Screening
9. Uncontrolled diabetes with an HbA1c > 8
10. Significant uncontrolled hypothyroidism (thyroid stimulating hormone [TSH] < 0.8 x lower limit of normal) with the exception of stably treated hypothyroidism and uncontrolled hyperthyroidism (thyroid stimulating hormone [TSH] < 0.8 x > 1.5 x upper Any other condition, disorder or finding which in the opinion of the investigator would adversely impact participant safety or the ability of the participant to complete the study, including compliance with all study requirements and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 weeks
  Range 0 to 25, higher score indicating more suicidal risk
Adverse Events Log | 6 weeks
  This log is cumulative and captures adverse events (including serious adverse events) of all participants throughout the study.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 | 6 weeks
  Scores range from 0 to 100 (where 0 = no disability; 100 = full disability).
Diagnostic Interview for Anxiety, Mood, and Obsessive-Compulsive and Related Neuropsychiatric Disorders (Self-report and Clinician Administered) | screening
  no score range
Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-SPQ) | screening
  no score range
Yale-Brown Obsessive-Compulsive Scale-Second Edition (Y-BOCS-II) Symptom Checklist and Severity Scale | 6 weeks
  Each item is rated from 0 (no symptoms) to 4 (extreme symptoms). A score of 0-7 is considered nonclinical. Scores ranging between 8 and 15 are considered mild. Scores between 16 and 23 are considered moderate and scores between 24-31 and 32-40 are considered severe and extreme, respectively.
Montgomery-Asberg Depression Scale (MADRS) | 6 weeks
  Total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression," 20 to 34 indicates "moderate depression," a score of 35 and greater indicates "severe depression," and a total score of 60 or greater indicates "very severe depression".
Hamilton Anxiety Rating Scale (HAM-A) | 6 weeks
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indi- cates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Clinician-Administered PTSD Scale for DSM-5 | 6 weeks
  Total severity score on the CAPS-5 represents the sum of the individual severity scores (0-4) for each of the 20 PTSD symptoms (CAPS-5 items 1-20 that have TR definite or probable). Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Brief Symptom Inventory (BSI) | 6 weeks
  Scores on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Higher scores indicate higher severity.
Difficulties in Emotion Regulation Scale (DERS) | From enrollment to the end of treatment at 6 weeks
  Responses ranging from 1 to 5, 36 items total. Higher scores indicate worse outcomes.
Southampton Mindfulness Questionnaire (SMQ) | From enrollment to the end of treatment at 6 weeks
  12 items are rated on a seven-point Likert scale, and the scores range from 0 to 72. Higher scores indicate better mindfulness outcomes.
Brief Experiential Avoidance Questionnaire (BEAQ) | From enrollment to the end of treatment at 6 weeks
  Scores range from 15 to 90, with higher scores indicating worse outcomes (greater experiential avoidance).
Self-Compassion Scale-Short Form (SCS-SF) | From enrollment to the end of treatment at 6 weeks
  Score range from 1 to 5, with higher scores indicating better outcomes (higher self-compassion).
Quality of Life Enjoyment & Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | From enrollment to the end of treatment at 6 weeks
  Scores range from 14 to 70, with higher scores indicating better outcomes.
Inventory for Depression and Anxiety Symptoms (IDAS-II) | From enrollment to the end of treatment at 6 weeks
  18 subscales each ranging from 1 to 90, higher scores indicating worse outcomes.
Ten-Item Personality Inventory (TIPI) | From enrollment to the end of treatment at 6 weeks
  The total personality score ranges from 10-70, with higher scores indicating more endorsement of the respective personality type.
Stanford Expectations of Treatment Scale (SETS) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 18, with higher scores indicating greater expectancy.
Mystical Experience Questionnaire (MEQ) | From enrollment to the end of treatment at 6 weeks
  Total score ranges from 0 to 150, with higher score indicating greater endorsement of mystical-type experience.
Psychological Insight Questionnaire (PIQ) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 5, with higher scores indicating more insight.
Challenging Experience Questionnaire (CEQ) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0-4 per sub scale, with higher scores indicating more challenging experience.
Ego Dissolution Inventory (EDI) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 100, with higher scores indicating more ego dissolution.
Emotional Breakthrough Inventory (EBI) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 100, with higher scores indicating more ego dissolution.
Theoretical Orientation Profile Scale-Revised (TOPS-R) | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 10, with higher scores indicating more endorsement of respective orientation.
Working Alliance Inventory-Short Revised (WAI-SR) | From enrollment to the end of treatment at 6 weeks
  Scores range from 15-60, with higher scores indicating higher alliance.
Alcohol Use Disorders Identification Test (AUDIT) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 40, with higher scores indicating worse outcomes.
Drug Use Disorders Identification Test (DUDIT) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 40, with higher scores indicating worse outcomes.
Fagerstrom Test for Nicotine Dependence (FTND) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 10, with higher scores indicating worse outcomes.
Persisting Effects Questionnaire (PEQ) | From enrollment to the end of treatment at 6 weeks
  Scores range varies depending on the sets of questions, with 143 total, with higher scores indicating more positive effect outcomes.
Psychedelic Integration Scale (PIS) | From enrollment to the end of treatment at 6 weeks
  Scores range from 1 to 5, with higher scores indicating better integration outcomes.
Dimensional Obsessive-Compulsive Scale (DOCS) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 80, with higher scores indicating worse outcomes.
Obsessive Beliefs Questionnaire-44 (OBQ-44) | From enrollment to the end of treatment at 6 weeks
  Scores range from 44 to 308, with higher scores indicating worse outcomes.
Beck Anxiety Inventory (BAI) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 63, with higher scores indicating worse outcomes.
Beck Depression Inventory (BDI-II) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 63, with higher scores indicating worse outcomes.
PTSD Checklist for DSM-5 (PCL) | From enrollment to the end of treatment at 6 weeks
  Scores range 0 to 80, with higher scores indicating worse outcomes.
Posttraumatic Maladaptive Beliefs (PMB) | From enrollment to the end of treatment at 6 weeks
  Scores range 15 to 105, with higher scores indicating worse outcomes.
daily diary | 7 consecutive days at night at the start of participation, daily between dosing and the 4- week follow-up,
  questions about daily events, stressors, mood, mind wandering, and rumination.
The Internal-External Locus of Control Short Scale-4 (IE-4) | From enrollment to the end of treatment at 6 weeks
  Locus of control is defined as a generalized expectation of internal or external control of reinforcement

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kelmendi, MD, Principal Investigator — Yale University; Gabrielle Agin-Liebes, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center - Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes